CLINICAL TRIAL: NCT05668117
Title: RFN-Advanced Retrograde Femoral Nailing System (RFNA) - Early Usage Case-Series Utilizing the Retrograde Femoral Nail-Advanced for Fixation and Stabilization of the Distal Femur and Femoral Shaft
Brief Title: RFN-Advanced Retrograde Femoral Nailing System
Acronym: RFNA
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Clay Spitler, Associate Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300008523
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-01

CONDITIONS: Femur Fracture
Keywords: Intramedullary Nail; Retrograde; Union
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Control: Historical patient data from other published studies in the literature
- Study participants: Adult patients with non-pathologic distal femur and femoral shaft fractures treated with the Depuy Synthes Advanced Retrograde femoral nail who had at least 6 months of follow up.
  Interventions: Device: Depuy Synthes Advanced Retrograde femoral nail

INTERVENTIONS:
Device: Depuy Synthes Advanced Retrograde femoral nail — The Advanced Retrograde Femoral Nailing System (RFNA) is designed to improve fixation and stabilization of distal femur and femoral shaft fractures by reducing toggle and loss of reduction.
  Groups: Study participants

SUMMARY:
This study is a retrospective chart review of the safety and performance Standard of Care data on individuals that have previously been implanted with the femur nail of the RFNA System for the internal fixation of the femur. Demographics, medical history, primary diagnosis, mechanism of injury, type of injury, clinical and radiographic evaluation of bone consolidation, and device-related adverse events were collected. Descriptive statistics were applied to the data collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years or older at the time of index procedure
2. Subjects who received the Depuy Synthes Advanced Retrograde Nail in accordance with the indications for use.
3. Subjects who have at least 6 months of follow-up.

Exclusion Criteria:

* Subject with less than 6 months of follow up, pathologic fractures, and patients < 18 years of age will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-pathologic distal femur and femoral shaft fractures treated with the Depuy Synthes Advanced Retrograde femoral nail.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Union | 6 months
  Rate of fracture union

SECONDARY OUTCOMES:
Infection | 6 months
  Rate of infection
Implant breakage | 6 months
  Rate of implant breakage
Implant removal | 6 months
  Rate of symptomatic implant removal
Malunion | 6 months
  Rate of malunion

CONTACTS AND LOCATIONS:
Overall Officials: Clay Spitler, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Ehlinger M, Ducrot G, Adam P, Bonnomet F. Distal femur fractures. Surgical techniques and a review of the literature. Orthop Traumatol Surg Res. 2013 May;99(3):353-60. doi: 10.1016/j.otsr.2012.10.014. Epub 2013 Mar 18. PMID 23518071
- [Background] Ricci WM, Gallagher B, Haidukewych GJ. Intramedullary nailing of femoral shaft fractures: current concepts. J Am Acad Orthop Surg. 2009 May;17(5):296-305. doi: 10.5435/00124635-200905000-00004. PMID 19411641
- [Background] Iannacone WM, Bennett FS, DeLong WG Jr, Born CT, Dalsey RM. Initial experience with the treatment of supracondylar femoral fractures using the supracondylar intramedullary nail: a preliminary report. J Orthop Trauma. 1994 Aug;8(4):322-7. doi: 10.1097/00005131-199408000-00008. PMID 7965294
- [Background] Ricci WM, Bellabarba C, Lewis R, Evanoff B, Herscovici D, Dipasquale T, Sanders R. Angular malalignment after intramedullary nailing of femoral shaft fractures. J Orthop Trauma. 2001 Feb;15(2):90-5. doi: 10.1097/00005131-200102000-00003. PMID 11232660
- [Background] Tucker MC, Schwappach JR, Leighton RK, Coupe K, Ricci WM. Results of femoral intramedullary nailing in patients who are obese versus those who are not obese: a prospective multicenter comparison study. J Orthop Trauma. 2007 Sep;21(8):523-9. doi: 10.1097/BOT.0b013e31813347ac. PMID 17805018
- [Background] Gregory P, DiCicco J, Karpik K, DiPasquale T, Herscovici D, Sanders R. Ipsilateral fractures of the femur and tibia: treatment with retrograde femoral nailing and unreamed tibial nailing. J Orthop Trauma. 1996;10(5):309-16. doi: 10.1097/00005131-199607000-00004. PMID 8814571
- [Background] Moed BR, Watson JT. Retrograde nailing of the femoral shaft. J Am Acad Orthop Surg. 1999 Jul-Aug;7(4):209-16. doi: 10.5435/00124635-199907000-00001. PMID 10434075
- [Background] Oh CW, Oh JK, Park BC, Jeon IH, Kyung HS, Kim SY, Park IH, Sohn OJ, Min WK. Retrograde nailing with subsequent screw fixation for ipsilateral femoral shaft and neck fractures. Arch Orthop Trauma Surg. 2006 Sep;126(7):448-53. doi: 10.1007/s00402-006-0161-2. Epub 2006 Jun 21. PMID 16810555
- [Background] Shah S, Desai P, Mounasamy V. Retrograde nailing of femoral fractures: a retrospective study. Eur J Orthop Surg Traumatol. 2015 Aug;25(6):1093-7. doi: 10.1007/s00590-015-1658-6. Epub 2015 Jul 1. PMID 26126587
- [Background] Jaarsma RL, Pakvis DF, Verdonschot N, Biert J, van Kampen A. Rotational malalignment after intramedullary nailing of femoral fractures. J Orthop Trauma. 2004 Aug;18(7):403-9. doi: 10.1097/00005131-200408000-00002. PMID 15289684
- [Background] El-Kawy S, Ansara S, Moftah A, Shalaby H, Varughese V. Retrograde femoral nailing in elderly patients with supracondylar fracture femur; is it the answer for a clinical problem? Int Orthop. 2007 Feb;31(1):83-6. doi: 10.1007/s00264-006-0137-4. Epub 2006 May 9. PMID 16683109
- [Background] Ricci WM, Bellabarba C, Evanoff B, Herscovici D, DiPasquale T, Sanders R. Retrograde versus antegrade nailing of femoral shaft fractures. J Orthop Trauma. 2001 Mar-Apr;15(3):161-9. doi: 10.1097/00005131-200103000-00003. PMID 11265005
- [Background] Singh SK, El-Gendy KA, Chikkamuniyappa C, Houshian S. The retrograde nail for distal femoral fractures in the elderly: high failure rate of the condyle screw and nut. Injury. 2006 Oct;37(10):1004-10. doi: 10.1016/j.injury.2006.01.005. Epub 2006 Feb 24. PMID 16499912